CLINICAL TRIAL: NCT05670223
Title: Healthy Activities Improve Lives
Acronym: HAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022P001782; R21AG067091 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2023-01-04 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Pilot Group (Experimental): Participants (N=30) will be recruited across two churches, MorningStar Baptist Church and People's Baptist Church, to examine the feasibility and acceptability of the HAIL Online platform. Participants will complete the 8-week F&S! exercise program (with access to the adjunct HAIL online platform), which will be delivered in-person as well as remote, and then continue to use the HAIL online platform during the 3-mo follow-up.
  Interventions: Other: Fit&Strong Exercise Program

INTERVENTIONS:
Other: Fit&Strong Exercise Program — The Fit and Strong! Program (F&S!) is an exercise program for older adults developed by a study consultant, Dr. Susan Hughes, with funding from the National Institute of Aging. It is tailored for the unique needs of older, underserved adults and targets modifiable factors depicted by the socioecological model is necessary. The F&S! exercise program assists older adults to improve strength and functioning.

SUMMARY:
The investigators have developed an online platform to support the 8-week, F&S! exercise program called the Healthy Activity Improves Lives (HAIL) online platform. The aims of this study are to conduct an open pilot trial with exit interviews (N=30) of the HAIL online platform in two racially diverse churches to evaluate its feasibility and acceptability (Hypothesis 1) as well as explore its efficacy (Hypothesis 2).

DETAILED DESCRIPTION:
This is an open pilot study to evaluate the feasibility and accessibility of the HAIL online platform. This study will enroll two cohorts (i.e., at two racially diverse churches) for a total number of 30 participants. This study will use a phone screen to assess participants' eligibility and explain the study procedures. Eligible individuals will then be given a link to complete an e-Consent in REDCap as well as instructions on how to access the HAIL online platform to complete assessments as part of the baseline visit. Participants will complete the 8-week F&S! exercise program (with access to the adjunct HAIL online platform), which will be delivered in-person as well as remote, and then continue to use the HAIL online platform during the 3-mo follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 60 years
* Participants are able to travel to one of the churches for the in-person F&S! exercise sessions
* Participants cannot be currently participating in a regular PA (physical activity) program (i.e., at least 100 min per week of moderate to vigorous physical activities)

Exclusion Criteria:

* Participants do not understand study procedures or are unable to participate in the verbal consent process
* Participants must have a physician responsible for their medical care
* Participants endorse an item on the Revised Physical Activity Readiness Questionnaire (rPAR-Q) as confirmed by their treating physician
* Participants who report any contraindication to exercising (e.g., recent ECG changes or myocardial infarction, unstable angina, uncontrolled arrhythmias, third degree heart block, congestive heart failure)

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and Retention | Week: 20
  Retention will be assessed by how many people completed the 3-month post-intervention follow-up
Acceptability | Week: 0
  Acceptability will be assessed by:1) Client Satisfaction Questionnaire (CSQ-8), 2) F&S! - online Feedback form, 3) Focus group exit interviews. The CSQ-8 assesses acceptability and feasibility of the F&S!-Online program and has demonstrated good reliability and validity.
  We will develop a form to ask for tailored feedback on the F&S-Online program to better understand participants' satisfaction with specific aspects of this online program.
  We will also conduct exit interviews with focus group and pilot study participants
Acceptability | Week: 8
  Acceptability will be assessed by:1) Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 assesses acceptability and feasibility of the F&S!-Online program and has demonstrated good reliability and validity.
Acceptability | Week: 20
  Acceptability will be assessed by :1) Client Satisfaction Questionnaire (CSQ-8), 2) F&S! - online Feedback form, 3) Focus group exit interviews. The CSQ-8 assesses acceptability and feasibility of the F&S!-Online program and has demonstrated good reliability and validity. We will develop a form to ask for tailored feedback on the F&S-Online program to better understand participants' satisfaction with specific aspects of this online program.
  We will also conduct exit interviews with focus group and pilot study participants

SECONDARY OUTCOMES:
Changes in Aerobic Capacity | Weeks: 0 , 8 , 20
  This outcome will be measured via the 6 minute Walk Test.
Changes in Physical Strength | Weeks: 0 , 8 , 20
  This outcome will be measured via the Timed-Stands Test.
Motivation to Change | Weeks: 0
  Motivation to change outcome will be measured via the Readiness for Change Form. This is used to measure participants' motivation to participate in exercising. A high score indicates the respondent is more interested in participating in exercise activities. A low score indicates the respondent is less interested in participating in exercise activities.
Utilization of Healthcare Resources | Weeks: 0
  Utilization of healthcare resources outcome will be assessed via the Healthcare Utilization Form. This a descriptive measure used to assess utilization of healthcare resources in the past 6 months, and to better characterize the sample based on the number of comorbid conditions present. There is no scoring or total score.
Fall History | Weeks: 0
  Fall history outcome will be measured via the Fall History Form. This form is used to assess the history of falling within the past two years in participants.
Chronic Conditions | Weeks: 0
  Chronic conditions outcome will be measured via the Geri-AIMS. This is a19-item self-administered questionnaire adapted from the Arthritis Impact Measurement Scales (AIMS) for use with frail elderly respondents. The questionnaire assesses the presence of existing chronic medical conditions.
Changes in Overall Wellbeing | Weeks: 0, 8 , 20
  Wellbeing will be measured via the WHO(Five) Well-Being Index (WHO-5). This is a reliable psychometric measure that predicts depression. The questionnaire consists of five items that assess predictors of depressive symptoms: positive mood, energy and interest. The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
Changes in Depression | Weeks: 0, 8 , 20
  Depression outcome will be measured via the Patient Health Questionnaire (PHQ-9). This is a 9-item, standardized and validated questionnaire that assesses the prevalence and severity of depression based on the DSM-5 criteria. The raw score ranges from 0 to 27, 1 representing minimal depression and 27 representing severe depression.
Changes in Anxiety | Weeks: 0, 8 , 20
  Anxiety outcome will be measured via the Generalized Anxiety Disorder 7-item (GAD-7) scale. This is a 7-item anxiety scale with good reliability, as well as criterion, construct, factorial, and procedural validity. The raw score ranges from 0 to 21. Increasing scores are associated with multiple domains of functional impairment. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Changes in Physical Functioning | Weeks: 0, 8 , 20
  Physical function outcome will be measured via the Patient-Reported Outcomes Measurement Information-Physical Functiong. This is an 8-item scale assessing coordination, functional mobility, strength and upper extremity function. The raw score ranges from 0 to 40. Increasing scores are associated with higher physical functioning.
Changes in Social Isolation | Weeks: 0, 8 , 20
  Social isolation outcome will be measured via the Patient-Reported Outcomes Measurement Information Short Form - Social Isolation 4. This is a 4-item scale used to capture participants' perception of being left out and disconnected from others. The raw score ranges from 0 to 20. Increasing scores are associated with higher feelings of social isolation.
Changes in Confidence in Exercises | Weeks: 0, 8 , 20
  Exercise confidence outcome will be measured via the Exercise Confidence Form. This is a 4-item questionnaire used to assess confidence in doing certain physical activities. The raw score ranges from 0 to 40. Increasing scores are associated with higher confidence in exercise.

OTHER OUTCOMES:
Satisfaction with program | Week: 8
  This outcome will be measured via the Client Satisfaction Questionnaire (CSQ-8). Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Satisfaction with program | Week: 20
  This outcome will be measured via the Client Satisfaction Questionnaire (CSQ-8). Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Use of online program | Weeks: 8
  This outcome will be assessed via the F&S! Program feedback from. This form consists of 8 questions and a semi-structured exit interview of 4 questions. There is no scoring or total score.
Use of online program | Weeks: 20
  This outcome will be assessed via the F&S! Program feedback from. This form consists of 8 questions and a semi-structured exit interview of 4 questions. There is no scoring or total score.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Sylvia, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States